CLINICAL TRIAL: NCT00014014
Title: A Phase I Pharmacokinetic Study of Once Versus Twice Daily Dosing With Zidovudine and Lamivudine
Brief Title: Zidovudine and Lamivudine Given Once Versus Twice Daily
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Model: Crossover | Purpose: Treatment
Other Study IDs: P1012; PACTG P1012; ACTG P1012; 11648 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2001-04-07; First posted 2001-08-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
Keywords: Zidovudine; Phosphorylation; Drug Administration Schedule; Lamivudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; Combivir
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination

INTERVENTIONS:
Drug: Lamivudine/Zidovudine

SUMMARY:
The purpose of this study is to see if the full daily dose of Combivir (zidovudine [ZDV]/lamivudine [3TC]) taken once a day is as effective as the usual recommended twice-a-day dose.

Studies have shown that the antiviral activity of ZDV can continue in the body even after there does not appear to be any ZDV left in the blood. This occurs because the body breaks down the drug into substances that remain active against HIV. The body also breaks down 3TC, a drug that is combined with ZDV in the Combivir product, in a similar way. Since antiviral activity may continue after Combivir is removed from the body, it may not be necessary to take the drug as often as once thought. This study carefully measures levels of the active substances in order to find out whether the same amount of antiviral activity occurs with less-frequent dosing.

DETAILED DESCRIPTION:
Initial dosing regimens of ZDV were based on the plasma half-life of the drug. However, recent studies of the intracellular metabolism of ZDV have demonstrated that the active anabolite, ZDV-TP, is present within the cell for an extended period of time relative to the drug in the plasma. This suggests that antiviral activity may be present for a sufficient time frame with less-frequent dosing of the drug. Careful comparison of the rate and extent of intracellular phosphorylated ZDV metabolites as a function of schedule will determine whether less-frequent dosing has a sound pharmacological basis. Also, the intracellular metabolism of 3TC is via different enzymes than that of ZDV and there are quantitative differences in the amount of triphosphate formed from both drugs. This study will provide information about intracellular metabolites when both ZDV and 3TC are concurrently administered.

This is a study of 2 schedules of Combivir therapy. At study entry or Part I, all patients take Combivir twice daily for the 7-day adherence assessment. Patients who have demonstrated 70 percent or greater adherence [AS PER AMENDMENT 7/20/01: 70 percent compliance with the study regimen for Combivir. This corresponds to taking at least 10 of the prescribed 14 Combivir tablets during the 7 days prior to an adherence assessment, including all scheduled doses in the 24-hour period prior to that assessment.], and have taken all scheduled Combivir doses in the previous 24 hours, have pharmacokinetic samples obtained and are randomized to Group A or Group B in Part II. Group A patients take 2 Combivir tablets once daily; Group B patients take 1 Combivir tablet twice daily. After patients have completed the targeted duration of Part II (7 days for Group A and 7-14 days for Group B), they are assessed for adherence. Patients who have demonstrated 70 percent or greater adherence, and have taken all scheduled Combivir doses in the previous 24 hours, have pharmacokinetic samples obtained and then change to the alternate dosing schedule. Group A patients take 1 Combivir tablet twice daily; Group B patients take 2 Combivir tablets once daily. After patients have completed the targeted duration of Part III (7-14 days for Group A and 7 days for Group B), they are assessed for adherence. All patients who meet the adherence criteria have pharmacokinetic samples obtained. After completion of Part III pharmacokinetic studies, patients have completed the study. (Note: Combivir will not be provided in this study.)

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 12 through 24 years of age.
* Are HIV-positive.
* Weigh more than 40 kg.
* Have a CD4 cell count above 250 cells/microL.
* Have taken at least 4 weeks of 3 or more anti-HIV medications, which must include ZDV and 3TC (as individual drugs or Combivir) and either a protease inhibitor or nonnucleoside reverse transcriptase inhibitor, and do not plan to change these medications during the study period.
* Have consent of a parent or guardian if under 18 years of age.
* Have a negative pregnancy test, if female and able to have children.
* Agree to use 2 effective methods of birth control (birth control pills plus a barrier method or 2 barrier methods) while taking study medication, if female and able to have children.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have an opportunistic (AIDS-related) infection that requires treatment at study entry.
* Are receiving anti-cancer medications for cancer.
* Are taking certain anti-HIV medications (nucleoside or nucleotide reverse transcriptase inhibitors, other than ZDV and 3TC), or hydroxyurea.
* Are pregnant or breast-feeding.
* Have diseases (other than HIV infection) or other conditions that, in the investigator's opinion, would interfere with the study.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, Study Chair
Locations (20):
- United States (19):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - St Joseph's Hosp & Med Center, Paterson, New Jersey
  - Metropolitan Hosp Ctr, New York, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
- Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan, Puerto Rico

REFERENCES:
- [Result] Flynn PM, Rodman J, Lindsey JC, Robbins B, Capparelli E, Knapp KM, Rodriguez JF, McNamara J, Serchuck L, Heckman B, Martinez J; PACTG P1012 Team. Intracellular pharmacokinetics of once versus twice daily zidovudine and lamivudine in adolescents. Antimicrob Agents Chemother. 2007 Oct;51(10):3516-22. doi: 10.1128/AAC.01626-06. Epub 2007 Jul 30. PMID 17664328